CLINICAL TRIAL: NCT05663840
Title: Progressive Resistance Exercise and Dystonia Pathophysiology.
Brief Title: Effects of Exercise on Dystonia Pathophysiology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202200490; 1R01NS122943 (NIH)
Record Dates: First submitted 2022-10-05; First posted 2022-12-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive resistance exercise (exercise group) (Experimental): Subjects will receive physical therapy that will predominantly include progressive resistance exercise training program along with continuation of standard of care (exercise group)
  Interventions: Behavioral: Progressive resistance exercise
- Standard of care (non-exercise group). (Active Comparator): Subjects will receive continuation of standard of care (non-exercise group).
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Progressive resistance exercise — Patients with predominant symptoms of cervical dystonia will receive exercise training. Patients will receive progressive resistance exercise focused cervical and shoulder training (PERFECT) plus standard-of-care (SOC) therapy. Resistance training will consist of mainly muscle-strengthening exercises for the neck, shoulder and arms and a few upper trunk muscles. Resistance training will be guided by physical therapists at twice a week schedule for 6 months. These participants will also receive SOC therapy.
  Arms: Progressive resistance exercise (exercise group)
Behavioral: Standard of care — Subjects will receive SOC therapy only
  Arms: Standard of care (non-exercise group).

SUMMARY:
The purpose of this research study is to investigate how the brain and motor behavior changes in individuals with dystonia in response to exercise training.

DETAILED DESCRIPTION:
Dystonia is a debilitating movement disorder. It involves involuntary muscle contractions with abnormal and repetitive movements, postures, or both. The current treatments for dystonia comprise of oral medications, botulinum toxin injections, and deep brain stimulation surgery. These treatments, despite optimal management, fail to improve symptoms in more than a third of patients and the improvements are often unpredictable. We will investigate the brain adaptation effects for progressive resistance exercise-focused cervical and shoulder training (PERFECT) in patients with focal cervical dystonia with functional MRI (fMRI) and transcranial magnetic stimulation (TMS) techniques for understanding the pathophysiology of dystonia and treatment related changes. The investigators propose to enroll patients with predominantly focal cervical dystonia and compare PERFECT plus standard-of-care (SOC) therapy (n = 27) with a control group of SOC therapy (n = 27). Participants in the PERFECT + SOC group will perform physical therapist-guided exercises twice a week for 6 months and participants in the SOC group will continue receiving standard pharmacological therapies at stable doses and they will not exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients have predominantly focal cervical dystonia and whose diagnosis will be confirmed by a movement disorders specialist following criteria recommended by Movement Disorders Society.
* Moderate disease severity.
* Are 30 to 85 years old
* Are able to tolerate exercise sessions.
* Reporting suboptimal clinical benefits despite receiving maximally tolerated doses of BoNT injections for the neck muscles and/or oral pharmacological therapy.

Exclusion Criteria:

* Participating in an alternate structured exercise program, receiving regular physical or occupational therapy
* Have significant pain, spondylosis or active arthritis
* Fail the Physical Activity Readiness Questionnaire
* Have significant cognitive impairment
* Have implanted electrical device (eg, cardiac pacemaker or a DBS or a neurostimulator or metallic clip in their body, as necessitated by the risks of MRI or TMS
* Active seizure disorder; not be eligible for TMS and claustrophobic for MRI portion. As necessitated by the risks of MRI or TMS, patients who have any type of implanted electrical device (such as a cardiac pacemaker or a neurostimulator), or a certain type of metallic clip in their body (i.e., an aneurysm clip in the brain), active seizure disorder are not eligible for participation in the MRI or TMS portion of the study.
* Pregnancy tests will be carried out for each female subject of child bearing potential prior to the participation in the study and prior to each follow up visit (as indicated).

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain effects measured with fMRI | Baseline up to 6 months
  To measure change in BOLD (fMRI) signals to functional connectivity in active group vs the control group.
Brain effects measured with TMS | Baseline up to 6 months
  To measure motor cortex excitability and plasticity in TMS findings.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle Shukla, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No